CLINICAL TRIAL: NCT00185081
Title: Radioimmunodetection of CEA-Producing Tumors Using a Bispecific Antibody Pre-targeting Method and an In-Labeled Peptide
Brief Title: Imaging Colo-rectal Cancer Using a Two Step Antibody Technique in Nuclear Imaging
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: PRISCO
Record Dates: First submitted 2005-09-15; First posted 2005-09-16 (Estimated); Last update posted 2016-04-07 (Estimated); Status verified 2016-04

CONDITIONS: Colonic Neoplasms
Keywords: colon cancer; radioimmunoscintigraphy; colon-specific antigen,; radioimmunotherapy,; radioimmunodetection
MeSH Terms: conditions — Colonic Neoplasms

INTERVENTIONS:
Drug: Indium labeled IMP-205xm734

SUMMARY:
The purpose of this study is to test the safety of the peptide and antibody and at the same time evaluate the tumor imaging of a two step antibody technique in nuclear imaging.

DETAILED DESCRIPTION:
Colo-rectal cancer has an incidence of 8000 cases per year in The Netherlands. Eventually 50% of them will die as a consequence of this disease.

Treatment consists of resection of the primary tumor, followed by adjuvant chemotherapy in some patients. The chemotherapeutical agents, however, are only moderately effective with regard to increase of survival. New treatment modalities are therefore desirable.

Radioimmunotherapy using radioactive labelled antibodies have proven to be effective in hematologic malignancies. Due to slow absorption in solid tumors however an effective radiation dose is not yet achieved.

The aim of our study is to bypass this slow tumor uptake by the use of pre-targeting. We therefore use an unlabeled bispecific antibody infusion. This will be followed several days later by the infusion of a radiolabeled peptide that binds to the bispecific antibody.

We hypothesise that this small peptide will be readily absorbed by the tumor which is pre-saturated by the bispecific antibody. As a consequence a higher radiation dose can be given with a lower toxicity.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years of age
* Histologic or cytologic diagnosis of colorectal cancer
* Karnofsky performance status >70%

Exclusion Criteria:

* Pregnant or lactating women
* Severe anorexia
* Active second primary malignancy
* Chemotherapy or radiotherapy within four weeks of study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2005-07; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Safety evaluation of intravenous injection of In-labeled IMP-205 and hMN-14xm734
Tumor targeting of In-IMP-205 in patients with colorectal carcinoma
Pharmacokinetics, biodistribution and dosimetry of In-IMP-205

CONTACTS AND LOCATIONS:
Overall Officials: Wim Oyen, MD PhD, Study Director — Radboud University Medical Centre Nijmegen
Locations (1):
- Radboud University Medical Centre Nijmegen, Nijmegen, Gelderland, Netherlands